CLINICAL TRIAL: NCT00035308
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Safety and Efficacy Trial of LJP 394 in Systemic Lupus Erythematosus (SLE) Patients With a History of Renal Disease
Brief Title: Safety and Efficacy Study of LJP 394 (Abetimus Sodium) to Treat Lupus Kidney Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: La Jolla Pharmaceutical Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LJP 394-90-09
Record Dates: First submitted 2002-05-02; First posted 2002-05-03 (Estimated); Last update posted 2006-09-25 (Estimated); Status verified 2002-12

CONDITIONS: Immunologic Diseases; Autoimmune Diseases; Systemic Lupus Erythematosus; Lupus Nephritis; Lupus Glomerulonephritis
Keywords: Immunologic Diseases; Autoimmune Diseases; Systemic Lupus Erythematosus; SLE; Lupus Nephritis; Lupus Glomerulonephritis
MeSH Terms: conditions — Immune System Diseases; Autoimmune Diseases; Lupus Erythematosus, Systemic; Lupus Nephritis | interventions — abetimus

INTERVENTIONS:
Drug: Abetimus sodium (LJP 394)

SUMMARY:
The purpose of this study is to determine whether LJP 394 (abetimus sodium) is safe and effective in delaying and reducing renal flares in patients with lupus nephritis.

DETAILED DESCRIPTION:
LJP 394 (abetimus sodium) is a unique drug that is specifically designed to lower production of antibodies to double-stranded DNA. These antibodies are believed to contribute to kidney damage in patients with Systemic Lupus Erythematosus (SLE). Rising levels of these antibodies seem to be associated with exacerbations of kidney disease that are known as "renal flares." Currently, anti-inflammatory and cytotoxic drugs are used to treat renal flares. Unfortunately, these drugs are often associated with certain unpleasant side effects. The purpose of this trial is to determine whether LJP 394 can delay or reduce the number of renal flares. It is possible that if renal flares can be delayed or reduced, patients may be able to take smaller amounts of anti-inflammatory or cytotoxic drugs and therefore suffer fewer of the side effects associated with these treatments.

ELIGIBILITY:
Inclusion Criteria

* Diagnosed with SLE
* Historical evidence of SLE renal disease
* Elevated levels of dsDNA antibodies
* Weight of 40 kg or greater

Exclusion Criteria

* Active SLE renal disease
* Use of certain anti-inflammatory or cytotoxic therapies or therapeutic interventions during the months immediately before dosing
* Clinical laboratory test values outside of certain limits
* Malignant disease or immunodeficiency syndrome
* Acute or chronic infections
* History of serious heart disease

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 330
Dates: Study Completion 2002-12

CONTACTS AND LOCATIONS:
Locations (82):
- United States (66):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Rheumatology Associates of North Alabama, Huntsville, Alabama
  - Montgomery Rheumatology Associates, Montgomery, Alabama
  - Arizona Arthritis & Rheumatology, Paradise Valley, Arizona
  - Allergy and Rheumatology Medical Clinic, La Jolla, California
  - Davida-USC Dialysis Center, Los Angeles, California
  - Wallace Rheumatic Study Center, Los Angeles, California
  - Private Practice, Los Angeles, California
  - UCLA School of Medicine, Los Angeles, California
  - Boling Clinical Trials, Rancho Cucamonga, California
  - Investigative Clinical Research, Rancho Cucamonga, California
  - Private Practice, San Mateo, California
  - Harbor-UCLA Research & Education Institute, Medicine/Rheumatology Division, Torrance, California
  - University of Connecticut Health Center, Division of Rheumatology, Farmington, Connecticut
  - Arthritis and Osteoporosis Center, PC, Hamden, Connecticut
  - CRIA Research, Fort Lauderdale, Florida
  - nTouch Research Corp., St. Petersburg, Florida
  - Emory University School of Medicine, Renal Division, Atlanta, Georgia
  - Private Practice, Macon, Georgia
  - Intermountain Research Center, Boise, Idaho
  - Radiant Research-Boise, Boise, Idaho
  - Northwestern University, Chicago, Illinois
  - Rheumatology Associates, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Rheumatology Consultants, Evansville, Indiana
  - Rheumatology Associates, PC, Indianapolis, Indiana
  - University of Louisville, Dept of Medicine/Division of Rheumatology, Louisville, Kentucky
  - LSU Health Sciences Center, Department of Rheumatology, New Orleans, Louisiana
  - Ochsner Clinic, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - SOMARC, Trials, LLC, Greenbelt, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Health System, Internal Medicine-Rheumatology, Ann Arbor, Michigan
  - Wayne State University, Rheumatology Division, Detroit, Michigan
  - Saint Louis University Health Sciences Center, St Louis, Missouri
  - Washington University, Renal Division, St Louis, Missouri
  - HIS Clinical Trials, Jersey City, New Jersey
  - SUNY-Downstate, Brooklyn, New York
  - Nephrology Associates, PC, Flushing, New York
  - NSUH-Division of Rheumatology, Manhasset, New York
  - Ambulatory Clinical Research Center, Hospital for Joint Diseases Orthopaedic Institute, NYU, New York, New York
  - Hospital for Joint Diseases, Department of Rheumatology, New York, New York
  - Hospital for Joint Diseases, NYU Medical Center, New York, New York
  - Mt. Sinai Medical Center, New York, New York
  - Columbia-Presbyterian Medical Center, New York, New York
  - AAIR Research Center, Rochester, New York
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Metrohealth Medical Center, Division of Rheumatology, Cleveland, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Oklahoma State University, Tulsa, Oklahoma
  - Healthcare Research Consultants, Tulsa, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Thomas Jefferson University, Division of Rheumatology, Philadelphia, Pennsylvania
  - University of Pittsburgh, Div. of Rheumatology and Clinical Immun., Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Dakota Regional Rheumatology, Rapid City, South Dakota
  - Medical Specialty Clinic, Jackson, Tennessee
  - University of Tennessee, Memphis, Memphis, Tennessee
  - Presbyterian Hospital of Dallas, Arthritis Consultation Center, Dallas, Texas
  - Radiant Research - Dallas, Dallas, Texas
  - Texas Tech University Health Sciences Center, Department of Internal Medicine, Lubbock, Texas
  - San Antonio Kidney Disease Center, Research Center, San Antonio, Texas
  - Clinical Research and Consulting Center, Fairfax, Virginia
  - MedSource, Inc., Richmond, Virginia
  - Arthritis Northwest, Spokane, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Division of Rheumatology, Department of Internal Medicine, Vienna, Austria
- Canada (2):
  - Arthritis Center of Excellence, Toronto Western Hospital, University Health Network, Toronto, Ontario
  - Hospital Maisonnueve-Rosemont, Montreal, Quebec
- Service De Rhumatologie Hopital de Hautepierre, Strasbourg, France
- Germany (3):
  - Universitatklinikum Charite, Medizinische Universitatsklinik, Berlin
  - MNR-Klinik/heinrich-Heine-University Dusseldorf, Düsseldorf
  - Department for Internal Medicine and Institute of Immunology and Rheumatology, Erlangen
- U.O di Reumatologia, Dipartimento di Medicina Interna, Universita di Pisa, Pisa, Italy
- Insituto Nacional de Ciencias Medicas Y Nutricion Salvador Zubiran, Depto. de Immunology y Rheumatology, Mexico City, Mexico
- Spain (3):
  - Hospital General Valle de Hebron Servicio Medicina Interna. Edificio, Barcelona
  - Hospital Clinic y Provinical de Barcelona, Unitat de Malalties Autoimmunes, Barcelona
  - Hospital Universitario La Paz Servico de Medicina, Madrid
- Sweden (2):
  - Department of Rheumatology, University Hospital of Lund, Lund
  - Department of Rheumatology, Karolinska Hospital, Stockholm
- United Kingdom (2):
  - Rheumatology and Rehabilitation Unit, Leeds
  - Lupus Research Unit St. Thomas Hospital, The Rayne Institute, London

REFERENCES:
- [Derived] Cardiel MH, Tumlin JA, Furie RA, Wallace DJ, Joh T, Linnik MD; LJP 394-90-09 Investigator Consortium. Abetimus sodium for renal flare in systemic lupus erythematosus: results of a randomized, controlled phase III trial. Arthritis Rheum. 2008 Aug;58(8):2470-80. doi: 10.1002/art.23673. PMID 18668592